CLINICAL TRIAL: NCT06054412
Title: Feasibility of an Adjunctive Dynamic Neurofeedback Training Program to Enhance Wellness Among Postpartum Mothers With a History of Trauma Exposure
Brief Title: An Adjunctive Neurofeedback Training Program to Enhance Wellness Among Trauma-Exposed Postpartum Mothers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Lisa S. Panisch, PhD, MSW, Assistant Professor, Wayne State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-23-02-5477
Record Dates: First submitted 2023-09-13; First posted 2023-09-26 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Well-Being, Psychological; Dissociation; Maternal Care Patterns; Maternal Behavior; Maternal Distress; Mood Disturbance; Emotional Regulation; Post Traumatic Stress Disorder
MeSH Terms: conditions — Psychological Well-Being; Dissociative Disorders; Emotional Regulation; Stress Disorders, Post-Traumatic | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neurofeedback Training (Other): Mothers in the Neurofeedback Training group will complete pre and post-training self-report surveys assessing trauma symptoms, mental health, parenting attitudes and behaviors, and infant crying patterns and socioemotional development. Mothers in this group will all be receiving in-person psychotherapy outside of the study, and they will all demonstrate clinically significant symptoms aligned with post-traumatic stress disorder and/or it's dissociative subtype.
  Interventions: Device: Neuroptimal (Zengar, Inc.) Neurofeedback

INTERVENTIONS:
Device: Neuroptimal (Zengar, Inc.) Neurofeedback — Mothers in the Neurofeedback Training group will complete one training session (lasting approximately 33 minutes) a week for a total of 12 weeks, using the Neuroptimal (Zengar, Inc.) neurofeedback device.

SUMMARY:
The proposed study will collect novel data evaluating the feasibility of the NFB training program delivered in an outpatient mental health setting and its influence on mothers' overall sense of well-being, and further investigate whether enhanced well-being is associated with positive changes in emotion regulation capacities, trauma-related mental health symptoms, parenting behaviors and attitudes, and infant behavioral outcomes (i.e., crying, fussing) among postpartum mothers with a history of childhood trauma and clinically concerning trauma-related mental health symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Must have clinically concerning symptoms of Post-traumatic Stress Disorder and/or it's dissociative sub-type, as indicated by either a score of 3+ on the Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) screening measure for PTSD symptoms OR endorsement of 2 or more past-month symptoms of moderate or greater severity on the depersonalization/derealization subscale of the Dissociative Subtype of PTSD Scale (DSPS).
* Must be between 3-24 months postpartum
* Must be receiving regular, primarily in-person psychotherapy from a therapist at a clinic in the Greater Detroit area.

Exclusion Criteria:

* Are currently pregnant
* Have a lifetime history of significant untreated mental illness (not currently treated schizophrenia, schizoaffective disorder, bipolar disorder, or substance use disorder) or neurological or pervasive developmental disorder
* Have a documented history of epilepsy
* Have ever experienced previous head injury with loss of consciousness
* Are currently experiencing domestic or intimate partner violence or otherwise state that their current living conditions are unsafe
* Are currently experiencing psychosis or have been suicidal within the last six months
* Are currently taking, or in the past month has taken benzodiazepines, narcotic drugs, or cannabis
* Have engaged in self-harming behaviors in the last 3 months requiring medical attention
* Do not have competence to understand or consent to the study procedures
* Do not have fluency in written and spoken English

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Neuro-QoL Item Bank v1.0 - Positive Affect and Well-Being - Short Form | Weekly, throughout the course of the 3-month training phase
  To measure maternal well-being. Minimum score = 9 Maximum score = 45 Higher scores mean a better outcome.
Post-Traumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders, Fith Edition (PTSD Checklist for DSM-5 - Standard) | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  To measure maternal symptoms of PTSD Minimum score = 0 Maximum score = 80 Higher scores mean a worse outcome.
Dissociative Experiences Scale II | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  To assess maternal symptoms of dissociation. Minimum score = 0 Maximum score = 100 Higher scores mean a worse outcome.
Patient Health Questionnaire 8 | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  To measure maternal depressive symptoms. Minimum score = 0 Maximum score = 24 Higher scores mean a worse outcome.
The State Trait Anger Expression Inventory | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  To measure maternal anger control. Minimum score = 10 Maximum score = 40 Higher scores mean a worse outcome.
Brief Child Abuse Potential screener, an abbreviated version of the Child Abuse Potential Inventory ([CAP]), © 1980, 1986, Joel S. Milner, PhD.) | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  The Brief Child Abuse Potential is a screening tool that is an abbreviated version of the Child Abuse Potential Inventory ([CAP]), © 1980, 1986, Joel S. Milner, PhD.). This measure is used to understand a caregiver's potential risk of perpetrating acts of child abuse. The measure includes 33 items; caregiver's endorse whether they "Agree" or "Disagree" with each item. Agree responses are given a score of 1, Disagree responses are given a score of 0.
  Minimum score = 0 Maximum score = 33 Higher scores mean a worse outcome.
Parenting Stress Index | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  To measure stress associated with parenting. Minimum score = 36 Maximum score = 180 Higher scores mean a better outcome.
Parenting Sense of Competence scale | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  To measure feelings of parental competency and self-efficacy. Minimum score = 0 Maximum score = 80 Higher scores mean a worse outcome.
The Crying Patterns Questionnaire | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  To measure infant crying and fussing patterns. Minimum score = 0 Maximum score = 80 Higher scores mean a worse outcome.
The Baby Pediatric Symptom Checklist of the Survey of Well-Being for Young Children | The measure will be administered at beginning of the study and again following the completion of the training phase, up to 4 months later.
  To measure infant psychosocial wellbeing. Minimum score = 0 Maximum score = 80 Higher scores mean a worse outcome.
Neuro-QoL Item Bank v1.0 - Emotional and Behavioral Dyscontrol - Short Form | Weekly, throughout the course of the 3-month intervention
  To measure maternal emotional and behavioral self-regulation. Minimum score = 0 Maximum score = 80 Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States